CLINICAL TRIAL: NCT04539834
Title: Electrolyte State in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Essamedin Mamdouh Negm, lecturer, Zagazig University
Other Study IDs: (ZU-IRB#: 6328-23-8-2020)
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Electrolyte Imbalance
Keywords: Electrolytes; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Electrolytes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: electrolytes — measuring level of electrolytes

SUMMARY:
Initial case reports and cohort studies have described many clinical characteristics of patients with coronavirus disease 2019 (COVID-19), an emerging infectious disorder caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). In early COVID-19 studies, some evidence has been provided that electrolyte disorders may also be present upon patients' presentation, including sodium, potassium, chloride and calcium abnormalities

the aim of the study is Identification of elements that affect COVID-19 pathology to improve survival and decrease mortality rate.

DETAILED DESCRIPTION:
SARS-CoV-2 invades human cells through binding angiotensin I converting enzyme 2 (ACE2) on the cell membrane. ACE2 is widely distributed in many types of human tissues, especially in the vital organs, such as heart, liver, kidney, and lungs. ACE2 is viewed as the principal counter-regulatory mechanism for the main axis of renin-angiotensin system (RAS) that is an essential player in the control of blood pressure and electrolyte balance. The final effect is to increase reabsorption of sodium and water, and thereafter increase blood pressure and excretion of potassium (K+). Besides, patients with COVID-19 often had gastrointestinal symptoms such as diarrhea and vomiting

Early studies proved that high percentage of COVID-19 patient were presented with electrolyte disorders, including sodium, potassium, chloride and calcium abnormalities. Such electrolyte disturbances have important implications not only for patient management but also for identifying potential pathophysiologic mechanisms underlying COVID-19 that could drive novel therapeutic opportunities

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old who were confirmed by the real-time PCR on the respiratory tract samples as positive of SARS-CoV-2.

Exclusion Criteria:

* Patients who had other causes of electrolyte disturbances (9):
* Chronic organ dysfunction (e.g., hepatic or renal dysfunction),
* Terminal cancer, immunodeficiency, and
* Patients with a history of long-term use of hormones & Diuretics were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old with diagnosis of COVID-19 infection who admitted to Isolation hospital of Zagazig University Hospitals during the period from 1 May 2020 to 1 August 2020.
Sampling Method: Probability Sample
Enrollment: 983 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
electrolytes disturbances in patients with COVID-19 | 4 months
  Serum Electrolytes (Na, K, Ca, Cl, Ph, Mg) abnormality in COVID 19 patients laboratory results in the different stages of the disease

SECONDARY OUTCOMES:
To asses the relation of the electrolyte disturbances with the severity of COVID-19 infection. | 4 months
  To find any correlation between the level of the electrolyte disturbances and the morbidity and mortality of the disease .

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Hamdy, MD, Study Director — lecturer of Chest diseases, Faculty of Medicine, Zagazig University; Hadeer El Shahaat, master degree, Principal Investigator — Assistant lecturer of Chest diseases, Faculty of Medicine, Zagazig University; Ahmed Abdulsaboor, MD, Principal Investigator — Clinical Pathology Department, Faculty of Medicine, Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt